CLINICAL TRIAL: NCT01172990
Title: Direct Angioplasty for Non ST Elevation Acute Coronary Events: DANCE Pilot Study
Acronym: DANCE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry); Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DANCE Pilot Study
Record Dates: First submitted 2010-07-26; First posted 2010-07-30 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Acute Coronary Syndrome
Keywords: ST Depression
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Group (Experimental): Patients allocated to the conventional management group will have medical stabilisation and will undergo angiogram +/- Percutaneous Coronary Intervention PCI between 24 to 48 hours from randomisation according to local policy and guidelines
  Interventions: Procedure: Conventional Management
- Immediate Invasive Group (Active Comparator): Patients allocated to the immediate invasive strategy will be taken to the catheter lab immediately (< 90 minutes from randomisation) in accordance with local primary angioplasty policy. Angiogram +/- same sitting Percutaneous Coronary Intervention(PCI) will be performed according to local policy and guidelines
  Interventions: Procedure: Immediate Invasive Management

INTERVENTIONS:
Procedure: Immediate Invasive Management — Patients allocated to the immediate invasive strategy will be taken to the catheter lab immediately (< 90 minutes from randomisation) in accordance with local primary angioplasty policy. Angiogram +/- same sitting PCI will be performed according to local policy and guidelines
  Arms: Immediate Invasive Group
Procedure: Conventional Management — Patients allocated to the conventional management group will have medical stabilisation and will undergo angiogram +/- PCI between 24 to 48 hours from randomisation according to local policy and guidelines
  Arms: Conventional Group

SUMMARY:
This is a pilot feasibility study to evaluate if patients with ST depression Acute Coronary Syndrome who are taken directly to the catheter laboratory for angiogram and angioplasty +/- stents will fare better that patients who are taken to the ward area and managed with drug therapy and stabilised for 24 hours before being taken to the catheter laboratory.

ELIGIBILITY:
Inclusion Criteria Patients presenting with symptoms (onset of symptoms ≤ 12 hours) of a suspected acute coronary syndrome (unstable angina or MI without persistent ST elevation) characterised as follows

* Clinical history consistent with ongoing ischaemic chest pain and/or symptoms AND
* >1mm ST depression AND/OR ≥2mm T wave inversion in at least two adjacent ECG leads Pathological T wave inversion in leads 1+4 suggesting 'LAD Syndrome' Or Ischaemic ST depression/T wave inversion not fulfilling the above criteria that is felt in the opinion of the attending physician to represent an acute coronary syndrome. AND
* Written informed consent Main exclusion criteria

  1. ≤ 18 years of age
  2. Previous Coronary Artery Bypass Grafting surgery
  3. ST elevation myocardial infarction
  4. Left bundle branch block (LBBB)
  5. ST depression seen in patients during paced mode only
  6. Heart rate ≥ 150bpm
  7. Cardiogenic shock or other catastrophic state
  8. If in the opinion of the physician the patient is not suitable for revascularisation due to co-morbidity
  9. Patient participating in another clinical trial such that randomisation to DANCE would result in deviation from the protocol stipulations of either trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Ambulance recruitment rate per million of population (corrected for 9-5 recruitment) | 12 months (duration of study)

SECONDARY OUTCOMES:
Percentage of patients recruited by the ambulance services ultimately manifesting a troponin positive Acute Coronary Syndrome(ACS) within 72 hours | within 72 hours
Percentage of ambulance recruited patients, excluded from the trial ultimately manifesting a troponin positive ACS within 72 hours | within 72 hours
The extent of myocardial damage will be evaluated using the area under the curve (AUC) for release of cardiac markers Creatinine Kinase Myocardial Band(CKMB) and troponin | within 7 days
Death at 30 days | at 30 days
Recurrent non-fatal Myocardial Infarction (MI) (after 72 hours) at 30 days | at 30 days
Additional unplanned revascularisation at 30 days. | at 30 days
Major bleeding | 30 days
Stroke at 30 days | at 30 days
Unplanned hospital stay (>72 hours) | within 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Miles Dalby, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton And Harefield NHS Trust, Harefield, Middlesex, United Kingdom